CLINICAL TRIAL: NCT01823757
Title: The Impacts of Pharmaceutical Cares on the Elderly in a VA Nursing Home.
Brief Title: Pharmaceutical Care in VA Nursing Home
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: VGHTCPHARMACY1; TCVGHPHARM_RESEARCH_1 (Other: Taichung Veteran General Hospital)
Record Dates: First submitted 2013-03-29; First posted 2013-04-04 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Focus on the Elderly in a Nursing Home
Keywords: elderly; potential inappropriate medications; pharmaceutical care; quality of life; medical expenditure
MeSH Terms: interventions — Pharmaceutical Services

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-pharmaceutical care: Veterans do not receiving pharmaceutical care
- Pharmaceutical care: Veterans receiving pharmaceutical care
  Interventions: Other: Pharmaceutical care

INTERVENTIONS:
Other: Pharmaceutical care — pharmacists provide pharmaceutical care to the intervention group, comparing to ordinary care in control group
  Groups: Pharmaceutical care

SUMMARY:
This study investigates the effect of pharmaceutical care on a Veteran nursing home. 100 patients will be selected into this controlled study.The hypothesis are:

1. After patients receive pharmaceutical care, their drug related problems will be decreased.
2. After patients received pharmaceutical care, their self-reported medical expenditure will be decreased.

DETAILED DESCRIPTION:
Around 200 residents in a Veteran nursing home will be selected for reviewing inclusion and exclusion criteria. A total of 100 subjected are selected into this randomized controlled trial. Each group will have 50 subjects and then divides into 4 subgroup, according to their drug items used (5-7 and over 8 items used).

The inclusion criteria:

1. Residents of the Veteran nursing home.
2. over 65 years old.
3. complete comprehensive geriatric assessment (CGA)
4. prescription drugs more than 4 times/day, excluding stat order.
5. with 2 or more chronic diseases.

Exclusion criteria:

1. residents who were in the pharmaceutical care project of Taiwan Pharmacists Association.

ELIGIBILITY:
Inclusion Criteria:

* Residents in the Veteran nursing home
* Age over 65 years old
* Complete Comprehensive Geriatric Assessment (CGA)
* Use more than 4 drug item per day (excluding stat order)
* subjects with more than 2 chronic diseases.

Exclusion Criteria:

* subjects who were in pharmaceutical care project of Taiwan Pharmacist Association.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Resident from a Veteran nursing home and willing to receive the pharmaceutical care by pharmacists.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
potential inappropriate medication (PIA) | one year

SECONDARY OUTCOMES:
drug items used | one year
  the controlled group is expected to have less drug items used.
medical expenditure | one year
  subjects self-reported outpatients visit, hospitalization, drug, and healthy supplemental used.

OTHER OUTCOMES:
quality of life measure | one year
  use health outcome measure, EQ-5D, to assess the quality of life issue.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Shyong Liou, PhD, Principal Investigator — Taichung Veteran General Hospital
Locations (1):
- Changhua Domiciliar Center, Changhua, Taiwan, Taiwan